CLINICAL TRIAL: NCT04993534
Title: RESPOND: Improving the Preparedness of Health Systems to Reduce Mental Health and Psychosocial Concerns Resulting From the COVID-19 Pandemic. A Randomized Controlled Trial in Italy
Brief Title: RESPOND: Improving the Preparedness of Health Systems to Reduce Mental Health and Psychosocial Concerns Resulting From the COVID-19 Pandemic
Acronym: RESPOND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universita di Verona (Other)
Collaborators: VU University of Amsterdam (Other); Universidad Autonoma de Madrid (Other); London School of Economics and Political Science (Other); Sorbonne University (Other); Mainz University (Other)
Responsible Party: Principal Investigator, Marianna Purgato, PhD, Assistant Professor, clinical psychologist, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 101016127
Record Dates: First submitted 2021-08-05; First posted 2021-08-06 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Psychological Distress
Keywords: mental health; psychological symptoms; resilience; wellbeing
MeSH Terms: conditions — Psychological Well-Being | interventions — Psychological First Aid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychological First Aid + Stepped-care intervention (DWM/PM+) (Experimental): All participants will be offered individual Psychological First Aid (PFA), a WHO developed support strategy that involves humane, supportive and practical help for individuals suffering from serious humanitarian crises.
  The treatment group will receive the stepped-care program consisting of DWM (step 1) and Problem Management Plus (PM+).
  The DWM program has been developed by WHO and collaborators working in the humanitarian field. DWM was designed to be relevant for large segments of adversity-affected populations: it is intended to be transdiagnostic, and easily adaptable to different cultures and languages.
  PM+ is a new, brief, psychological intervention program based on cognitive-behavioral therapy (CBT) techniques that are empirically supported.
  Interventions: Behavioral: Stepped-care DWM/PM+
- Psychological First Aid + usual care (Other): All participants will be offered individual Psychological First Aid (PFA), a WHO developed support strategy that involves humane, supportive and practical help for individuals suffering from serious humanitarian crises.
  In addition, both the groups will receive care-as-usual (CAU); they will be allowed to receive any usual care. CAU may include community care, social/legal support, and psychoeducation.
  Interventions: Other: Psychological First Aid + usual care (CAU)

INTERVENTIONS:
Behavioral: Stepped-care DWM/PM+ — The DWM program consists of a self-help guide that is complemented with pre-recorded audio exercises. The audio material imparts key information about stress management and guides participants through individual exercises. Additionally, participants are guided by a briefly trained helper. DWM includes five sections (or modules), each of which focuses on a specific skill. In this study, the DWM program will be delivered as an online intervention. The DWM intervention, i.e. both the audios and the self-help guide, have been adapted for use on a smartphone or other device with internet access.
  PM+ is a new, brief, psychological intervention program based on cognitive-behavioral therapy (CBT) techniques. The manual involves the following empirically supported elements: problem solving plus stress management, behavioral activation, facing fears, and accessing social support.
  Arms: Psychological First Aid + Stepped-care intervention (DWM/PM+)
Other: Psychological First Aid + usual care (CAU) — All participants, both in the treatment and the comparison group, will be offered individual Psychological First Aid (PFA) through a face-to-face or teleconferencing meeting. In addition to PFA, both the treatment and the comparison group will receive care-as-usual (CAU); they will be allowed to receive any usual care. CAU may include community care, social/legal support, and psychoeducation.
  Arms: Psychological First Aid + usual care

SUMMARY:
This randomized controlled trial will evaluate the implementation and (cost-)effectiveness of the culturally and contextually adapted Doing What Matters in times of stress (DWM) and Problem Management Plus (PM+) stepped-care programs amongst asylum seekers, refugees, and/or migrants living in Italy. Outcomes include mental health, resilience, wellbeing, health inequalities, and costs to health systems.

DETAILED DESCRIPTION:
Rationale: The ongoing COVID-19 pandemic has a major and potentially long-lasting effect on mental health and wellbeing across populations worldwide. Vulnerable groups, such as asylum seekers, refugees and migrants, are disproportionally affected by the COVID-19 pandemic. There is a high need for psychosocial interventions that can target the most prevalent mental health problems as a result of the COVID-19 pandemic, addressing the needs of many people in a way that maximizes the use of resources. The World Health Organization (WHO) has developed two scalable, low-intensity psychological interventions: Doing What Matters in times of stress (DWM; a self-help intervention) and Problem Management Plus (PM+; a face-to-face intervention). DWM and PM+ can be delivered by paraprofessionals, are applicable to a variety of mental health problems (depression, anxiety and PTSD), and can be adapted to different populations, cultures and languages. Both DWM and PM+ have been proven to be effective on their own. In this study, DWM and PM+ will be combined into a stepped-care intervention. This study is part of the larger EU H2020-RESPOND project, which aims to improve the preparedness of the European mental health care system in the face of future pandemics.

Objective: The main objective is to evaluate the implementation and (cost-)effectiveness of the culturally and contextually adapted DWM/PM+ stepped-care programs amongst asylum seekers, refugees, and/or migrants living in Italy during the COVID-19 pandemic in terms of mental health outcomes, resilience, wellbeing, health inequalities, and costs to health systems. The main hypothesis is that the stepped-care DWM/PM+ intervention together with psychological first aid (PFA) in addition to care-as-usual (CAU) will be more effective in decreasing psychological distress and symptoms of mental health problems than PFA and CAU alone. We aim to conduct a randomized controlled trial (RCT) to assess the (cost-)effectiveness of the stepped-care DWM/PM+ intervention, and to identify (a) barriers and facilitators to treatment engagement and adherence and (b) opportunities for scaling up the implementation of the DWM/PM+ intervention within the existing health care system in Italy.

Study design: pragmatic implementation trial with a single-blinded, randomized, parallel-group design. The final phase of the trial will consist of a qualitative process evaluation with individual interviews and focus group discussions (FGDs).

The qualitative phase will include some participants in the randomized trial who completed DWM (n=2/4;), who completed PM+ (n=2/4), who dropped-out during DWM (n=2/4), and who dropped-out during PM+ (n=2/4); (b) local stakeholders (n=10/15) (c) facilitators of the DWM and PM+ intervention (both helpers and trainers/supervisors).

Study population: Adult asylum seekers, refugees or migrants with self-reported elevated psychological distress (K10 >15.9) (n=212).

Intervention: All participants (in both the treatment and the comparison group) will receive Psychological First Aid (PFA) and CAU. In addition to PFA and CAU, the treatment group will receive the stepped-care intervention (DWM with or without PM+). The stepped-care intervention consists of DWM (step 1), and conditionally PM+ (step 2) if participants still meet criteria for psychological distress (K10 >15.9) 2 weeks after having received DWM.

DWM, i.e. a self-help book with pre-recorded audios, has been adapted as an online intervention (phase 1). PM+ consists of five sessions and will be delivered by trained peer-support helpers in person or via teleconferencing in individual or group format. In addition to PFA, the comparison group will receive CAU which ranges from community care to specialized psychological treatments, according to the needs and clinical characteristics of participants.

Main study parameters/endpoints: Screening for inclusion and exclusion criteria will be interviewer-administered, inperson or through (video) calls. For all participants, online assessments will take place at baseline, at 2 weeks after having received DWM, at 1 week and at 2 months after having received PM+. The primary outcome will be the decrease in symptoms of anxiety and depression from baseline to two-month follow-up, measured through the sum score of the Patient Health Questionnaire (PHQ-9) and General Anxiety Disorder-7 (GAD-7), i.e. the PHQ-Anxiety and Depression Score (PHQ-ADS). We expect to detect a Cohen's d effect size of 0.3 in the DWM/PM+ group at 2 months post-treatment. Additional health outcomes include level of anxiety (GAD-7) and depression (PHQ-9), symptoms of posttraumatic stress disorder (PCL-5), resilience (Mainz Inventory of Microstressors, MIMIS), quality of life (5-level EQ-5D version, EQ-5D-5L), and cost of care (Client Service Receipt Inventory, CSRI). Additional study parameters will include demographic data, COVID-19 related (exposure) variables, treatment fidelity, satisfaction and acceptability of the intervention program, and implementation indicators (such as reach, dose, resource use, intervention-related costs). Through FGDs and interviews at the end of the trial, the feasibility of scaling-up the implementation on the stepped-care DWM/PM+ intervention within asylum seekers, refugees, and migrants in Italy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* Living in Italy as asylum seeker, refugee, or migrant
* Having elevated levels of psychological distress (Kessler Psychological Distress Scale (K10) >15.9).
* Sufficient mastery (written and spoken) of one of the languages the DWM/PM+ intervention is being delivered in (e.g. English, Italian).
* Oral and written informed consent before entering the study.

Exclusion Criteria:

* Planning to permanently move back to their home country before the last quantitative assessment at 2 months after PM+;
* Having acute medical conditions (requiring hospitalization);
* Imminent suicide risk, or expressed acute needs or protection risks that require immediate follow-up;
* Having a severe mental disorder (e.g. psychotic disorders, substance-dependence);
* Having severe cognitive impairment (e.g. severe intellectual disability or dementia);
* Currently receiving specialized psychological treatment (e.g. Eye Movement Desensitization and Reprocessing - EMDR; Cognitive behavioural therapy - CBT);
* In case of current psychotropic medication use: being on an unstable dose for at least 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire - Anxiety and Depression (PHQ-ADS) | Two-month follow-up after the PM+ intervention ended
  Decrease in symptoms of depression and anxiety. The total score ranges from 0 to 48, with higher scores indicating higher levels of depression and anxiety symptomatology.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | T1 (baseline), T2 (up to 2 weeks after DWM), T3 (up to 2 weeks after PM+), T4 (2 months after PM+)
  Level of depression The total score ranges from 0 to 27, with higher scores indicating higher levels of depression symptomatology.
Generalized Anxiety Disorder checklist (GAD-7) | T1 (baseline), T2 (up to 2 weeks after DWM), T3 (up to 2 weeks after PM+), T4 (2 months after PM+)
  Level of anxiety The total score ranges from 0 to 21, with higher scores indicating higher levels of anxiety symptomatology.
PTSD Checklist for DSM-5 (PCL-5) | T1 (baseline), T2 (up to 2 weeks after DWM), T3 (up to 2 weeks after PM+), T4 (2 months after PM+)
  Severity of posttraumatic stress disorder The total score ranges from 0 to 32, with higher scores indicating higher levels of PTSD symptomatology.
EuroQol five dimension five level checklist for quality of life EU European Union (EQ-5D-5L) | T1 (baseline), T2 (up to 2 weeks after DWM), T3 (up to 2 weeks after PM+), T4 (2 months after PM+)
  Quality of life
Mainz Inventory of MIcrostressorS (MIMIS) and stressful events | T1 (baseline), T2 (up to 2 weeks after DWM), T3 (up to 2 weeks after PM+), T4 (2 months after PM+)
  Resilience based on exposure to stressful (general- and COVID-19 related-) events (MIMIS)
Client Service Receipt Inventory (CSRI) | T1 (baseline), T2 (up to 2 weeks after DWM), T3 (up to 2 weeks after PM+), T4 (2 months after PM+)
  Cost of care: impact on use of health system, other services, time out of employment and other usual activities and need for informal care

CONTACTS AND LOCATIONS:
Locations (1):
- Università di Verona, Verona, VR, Italy

REFERENCES:
- [Derived] Purgato M, Turrini G, Tedeschi F, Serra R, Tarsitani L, Compri B, Muriago G, Cadorin C, Ostuzzi G, Nicaise P, Lorant V, Sijbrandij M, Witteveen AB, Ayuso-Mateos JL, Mediavilla R, Haro JM, Felez-Nobrega M, Figueiredo N, Pollice G, McDaid D, Park AL, Kalisch R, Petri-Romao P, Underhill J, Bryant RA, Nose M, Barbui C. Effectiveness of a stepped-care programme of WHO psychological interventions in migrant populations resettled in Italy: Study protocol for the RESPOND randomized controlled trial. Front Public Health. 2023 Jan 25;11:1100546. doi: 10.3389/fpubh.2023.1100546. eCollection 2023. PMID 36761135

DOCUMENTS (1):
  • Study Protocol (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT04993534/Prot_001.pdf